CLINICAL TRIAL: NCT03817034
Title: Multimodal Analgesia for the Reduction of Postoperative Opioid Consumption
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: We decided to close this study and come up with a new study design.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Emery Brown, Director, Neuroscience Statistics Research Laboratory, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018P002053
Record Dates: First submitted 2018-11-23; First posted 2019-01-25 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Pain
Keywords: multimodal; dexmedetomidine; ropivacaine; ketorolac; pain management; opioid sparing; analgesia
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Multimodal Analgesia (Experimental)
  Interventions: Drug: Multimodal analgesia

INTERVENTIONS:
Drug: Multimodal analgesia — Subjects will be given a rectus sheath block containing dexmedetomidine, ropivacaine, and ketorolac

SUMMARY:
The investigators are performing this research study to investigate the efficacy of local infiltration of the surgical wound combining dexmedetomidine, ropivacaine, and ketorolac (treatment group) versus the current standard of care (historical control group), for post-operative pain management.

DETAILED DESCRIPTION:
During this research study, patients recommended for a rectus sheath block during surgery will receive a novel combination of non-opioid drugs. Data from the treatment group will be compared to surgical outcomes of a historically matched control group to investigate the ability of this drug combination to reduce post-operative pain and post-operative opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* American Society of Anesthesiologist Physical Status Classification 1-3
* Undergoing surgery requiring a rectus sheath block

Exclusion Criteria:

* American Society of Anesthesiologist Physical Status Classification of 4 or beyond
* history of opiate of illicit substance abuse, chronic pain, or neurological dysfunction

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2021-03-11 (Actual)

PRIMARY OUTCOMES:
Change in post-operative opioid consumption | 48 hours
  Decreased post-operative opioid consumption associated with use of multimodal analgesia
Change in post-operative pain scores | 48 hours
  Decreased post-operative pain scores associated with use of multimodal analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Emery N Brown, M.D., Ph.D., Principal Investigator — Massachusetts General Hospital